CLINICAL TRIAL: NCT01494831
Title: Evaluation of a Group-based, Cognitive-behavioural Intervention With Former Child Soldiers and Other War-affected Children in the Democratic Republic of Congo: A Randomised Controlled Trial.
Brief Title: Randomized Control Trial of Group Intervention With Former War-affected Boys in the Democratic Republic of Congo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, John McMullen, Principal Investigator, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PREC23
Record Dates: First submitted 2011-12-15; First posted 2011-12-19 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Post-traumatic Stress Disorder; Depression; Conduct Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Conduct Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TF-CBT (Experimental)
  Interventions: Behavioral: TF-CBT
- Waiting List control (No Intervention)

INTERVENTIONS:
Behavioral: TF-CBT — 15 sessions of group-based, trauma-focused cognitive behavioral therapy
  Other Names: Trauma-focused Cognitive Behavioral Therapy
  Arms: TF-CBT

SUMMARY:
The purpose of this study is to evaluate, in a randomised control trial (RCT), the effectiveness of group-based, trauma-focused Cognitive Behaviour Therapy (TF-CBT) in reducing psychological distress in former child soldiers and other war-affected children in the Democratic Republic of Congo (DRC).

DETAILED DESCRIPTION:
To the best of the author's knowledge this is the first group-based mental health or psychosocial intervention developed specifically for psychologically distressed former child soldiers. While CBT is the modality with most empirical evidence for treating war-affected young people, this is the first evaluation with child soldiers specifically.

Former child soldiers and war affected 'street boys' (aged 13-17) in eastern DRC, will be screened for symptoms of psychological distress and then randomly assigned to either a treatment group or a waiting-list control. The treatment groups will receive a 15-session manualised, culturally-adapted, TF-CBT intervention. This includes psycho-education, relaxation, affect modulation, cognitive processing and constructing a trauma narrative. After treatment and post-testing, the waiting-list controls then begin their intervention.

ELIGIBILITY:
Inclusion Criteria:

* War-affected children and adolescents

Exclusion Criteria:

* No traumatic war events experienced
* Psychosis
* Inability to speak Swahili, French or English

Ages: 13 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2011-05; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Change in post-traumatic stress symptoms measured by UCLA-PTSD-RI | Post-intervention and 3 month

SECONDARY OUTCOMES:
Change in psychosocial distress- measures by African Youth Psychosocial Assessment | Post-intervention and 3 month
  Psychosocial distress- depression, anxiety, conduct problems, antisocial behaviour

CONTACTS AND LOCATIONS:
Overall Officials: Harry Dr Rafferty, Study Director — Queens University Belfast

REFERENCES:
- [Derived] McMullen J, O'Callaghan P, Shannon C, Black A, Eakin J. Group trauma-focused cognitive-behavioural therapy with former child soldiers and other war-affected boys in the DR Congo: a randomised controlled trial. J Child Psychol Psychiatry. 2013 Nov;54(11):1231-41. doi: 10.1111/jcpp.12094. Epub 2013 Jun 6. PMID 23738530